CLINICAL TRIAL: NCT05534815
Title: Long-Term Treatment of Opioid Use Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Michigan University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00325677; R01DA053218-01A1 (NIH)
Record Dates: First submitted 2022-09-06; First posted 2022-09-10 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Drug Addiction; Employment
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Usual Care Control group (No Intervention): Participants in the Usual Care Control group will receive methadone or buprenorphine treatment, counseling, and employment services.
- Initiation Only group (Experimental): Participants assigned to the Initiation Only group will be able to earn abstinence-contingent stipends for working with the employment specialist for up to 20 hours per week and performance stipends for engaging in job-seeking behaviors. When employed, those participants will be able to earn abstinence-contingent wage supplements for up to 40 hours worked (verified by pay stubs) in a community job. Participants can earn from both Therapeutic Workplace Work Hours and from wage supplements for working in a community job, however, participants will only be able to earn stipends and wage supplements for a maximum total of 40 hours.
  Interventions: Behavioral: Employment-based abstinence reinforcement
- Initiation and Maintenance group (Experimental): The Initiation and Maintenance group procedures will receive the same intervention as the Initiation Only participants for 24 weeks (during the Initiation period). Then, Initiation and Maintenance participants will receive a low-magnitude incentive intervention for 24 weeks (the Maintenance period, weeks 25-48) to maintain drug abstinence and employment. The low-magnitude incentive intervention will be identical to the final weeks of the high magnitude incentive intervention, with two important exceptions.
  1. During the low-magnitude intervention, participants will receive money per hour for maintaining drug abstinence and work (stipends for working with the employment specialist and wage supplements for providing pay stubs).
  2. During weeks 25-48, if a participant in the Initiation and Maintenance group provides a drug-positive urine sample or misses a required mandatory sample, the participant will not receive any incentive.
  Interventions: Behavioral: Employment-based abstinence reinforcement

INTERVENTIONS:
Behavioral: Employment-based abstinence reinforcement — Participants will earn stipends for working with the employment specialist and wage supplements for working in a community job, but the stipends and wage supplements will depend on providing drug-free urine samples.
  Arms: Initiation Only group; Initiation and Maintenance group

SUMMARY:
Poverty and opioid addiction are interrelated and chronic problems which have not been addressed adequately. The Therapeutic Workplace could treat the many adults with opioid use disorder who are unemployed and live in poverty. The Therapeutic Workplace pays participants to work. To promote drug abstinence, the Therapeutic Workplace arranges employment-based abstinence reinforcement in which participants are required to provide drug-free urine samples to maintain maximum wages. Many studies have shown that employment-based abstinence reinforcement in the Therapeutic Workplace can promote and maintain drug abstinence. Recently, the investigators showed that abstinence-contingent wage supplements in the Therapeutic Workplace could promote drug abstinence and employment and reduce poverty. However, the investigators have not demonstrated the real-world impacts of the Therapeutic Workplace. The Therapeutic Workplace requires two modifications to produce real world impacts.

1. The investigators must develop a real-world version of the Therapeutic Workplace that community treatment programs can implement.
2. The investigators must reduce the costs of maintaining employment-based abstinence reinforcement.

This application seeks to develop and evaluate a low-cost Therapeutic Workplace that community treatment programs can implement and that addresses the persistent nature of opioid addiction and poverty. The investigators propose to conduct a Stage III study in which a community clinic (REACH Health Services) adapts and implements the Therapeutic Workplace intervention. To improve the feasibility of this intervention, the investigators will use low-cost abstinence-contingent wage supplements to maintain abstinence. The investigators propose to conduct a randomized controlled study to evaluate the effectiveness of the low-cost abstinence-contingent wage supplements in a community Therapeutic Workplace to maintain long-term drug abstinence and employment, and to reduce poverty in adults with opioid use disorder. All participants will be invited to attend a 4-week induction period and 48 weeks of support by an employment specialist. At the end of a 4-week induction period, REACH unemployed methadone or buprenorphine patients with opioid use disorder who meet the Induction Period inclusion criteria (N=225) will be randomly assigned to a "Usual Care Control," an "Initiation Only," or an "Initiation and Maintenance" group. All groups will be offered methadone or buprenorphine treatment and an employment specialist for 48 weeks. "Initiation Only" and "Initiation and Maintenance" participants will earn high magnitude abstinence-contingent wage supplements during a 24-week Initiation period (weeks 1-24). "Initiation and Maintenance" participants will also earn low-magnitude abstinence-contingent wage supplements during a 24-week Maintenance period (weeks 25-48). The investigators will base the primary outcome measures on assessments conducted every four weeks of the Maintenance period. If low-cost abstinence-contingent wage supplements in the community Therapeutic Workplace maintain drug abstinence and employment and decrease poverty, community drug abuse treatment clinics could apply this intervention widely as a long-term maintenance treatment for unemployed adults with opioid use disorder.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* are enrolled at REACH for buprenorphine or methadone maintenance treatment
* unemployed

Exclusion Criteria:

* Applicants will be excluded if they report recent hallucinations and if they are currently a prisoner.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2028-02-29 (Estimated)

PRIMARY OUTCOMES:
Rate of Drug abstinence as assessed by a yes or no | 4 weeks
  We will assess rate of urine samples negative for opioids (morphine, oxycodone, and fentanyl) and cocaine at the 4-week assessments during the Maintenance period. Y/N at each assessment).
Rate of Employment as assessed by a yes or no | 4 weeks
  We will assess rate that participants report employment at the 4-week assessments conducted during the Maintenance period. Y/N at each assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Forrest Toegel, PhD, Principal Investigator — Northern Michigan University
Locations (1):
- Northern Center for Learning and Health, Northern Michigan University, 1401 Presque Isle Ave., Marquette, Michigan, United States

IPD SHARING:
Plan to Share IPD: No